CLINICAL TRIAL: NCT03881137
Title: Improving Function and Quality of Life for Older Cancer Patients Receiving Radiotherapy, a Randomized Controlled Pilot Study
Brief Title: Improved Function and Quality of Life for Older Patients Receiving Radiotherapy, Part II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sykehuset Innlandet HF (Other)
Collaborators: Trondheim University Hospital (Other); Norwegian University of Science and Technology (Other); Trondheim Kommune (Other); Oslo University Hospital (Other); University of Oslo (Other); Oslo Metropolitan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SI0303150406
Record Dates: First submitted 2019-03-13; First posted 2019-03-19 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Cancer; Radiotherapy; Older Patients
Keywords: older; cancer; radiotherapy; geriatric assessment; quality of life; physical function
MeSH Terms: conditions — Neoplasms | interventions — Geriatric Assessment; Therapeutics

STUDY DESIGN:
Intervention Model Description: The present study is a controlled cluster-randomized pilot study. Cluster-randomization is chosen to avoid contamination of the control group. Before patient recruitment commences, a selection of 32 municipalities and city districts (= clusters) will be stratified into blocks in accordance with number of inhabitants. The selection will include city districts, large and smaller municipalities to ensure sample size and representativity. Clusters within each block will be randomly assigned to intervention or control by using a computer-generated code, 1:1, i.e. 16 in each group
  Eligible, consenting patients from municipalities/city districts randomized to control will enter the control group. Eligible, consenting patients from municipalities randomized to intervention will enter the intervention group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Geriatric assessment with management
  Interventions: Other: Geriatric assessment with management
- Control (No Intervention): Patients receiving supportive care and follow up according to routine practice

INTERVENTIONS:
Other: Geriatric assessment with management — A multicomponent intervention, carried out in cooperation between hospital and community services, based on a geriatric assessment (GA) followed by individually adapted measures targeting identified needs.
  The GA and the start of the intervention will be handled by a PhD student (geriatrician) or project cancer nurse at start of RT. Pre-planned guidelines will be followed. Contribution from relevant hospital professionals will be sought according to needs. Then the intervention will be offered in the primary health care taking advantage of existing services, e.g. home care, rehabilitation services, exercise groups etc. A community-based coordinating nurse will follow the patients with weekly contacts throughout RT and to end of intervention 8 weeks post-RT. To ensure that each patient's intervention is properly adjusted to changing needs, repeated clinical assessments will be performed by the end of RT and 4 weeks post-RT.
  Arms: Intervention

SUMMARY:
This cluster randomized controlled pilot study is designed to test the feasibility, and potential effect of a multicomponent, community-based intervention aiming to improve quality of life (QoL) and function for older patients receiving radiotherapy (RT), and thereby reduce the needs for professional help. The intervention will be based on geriatric assessment and management (GAM), i.e. systematic assessment and management of physical, mental and functional problems frequently occurring in the elderly. It will target individual patients according to needs and be carried out in collaboration between hospital and community services from start of RT until 8 weeks post-treatment.

DETAILED DESCRIPTION:
Background:

Older cancer patients (> 65 years) represent the majority of the cancer population, and their number grows due to an aging population. These patients often present with a multiplicity of problems. They frequently suffer from physical- or mental health comorbidities, and are often frail with impairment in mobility, daily life functioning and cognition. When diagnosed with cancer and in need of therapy, they are at substantial risk of complications and functional decline.

Geriatric assessment with management (GAM) has documented success in improving outcomes in older patients with other diseases than cancer. Thus, GAM is strongly recommended as an approach to optimize treatment and care for older cancer patients. Evidence for the potential benefits is still scarce and in particular for older patients receiving radiotherapy.

Although GAM has been proven successful in other contexts, there is no universally accepted recipe for how such an intervention should be performed and implemented. To be feasible and efficient, adjustments according to patient population, health care organization and available resources are necessary. The present study will be conducted to provide the evidence needed for a subsequent definitive evaluation of a GAM intervention for older patients receiving radiotherapy in a larger RTC, aiming at improving quality of life (QoL) and function, and thereby reduce the burden for the patients, their families and the society.

The detailed objectives are to:

1. assess the potential short- and long-term effect of the intervention on global QoL and physical functioning for older cancer patients receiving RT
2. assess the feasibility of the intervention

   1. at the patient level (recruitment, compliance and adherence)
   2. at the organizational level (structures facilitating or impeding implementation and collaboration across sectors and between professionals)
3. study the use of health care services and related costs in the intervention and control group

Methods:

The study emerges from Innlandet Hospital Trust and will be conducted in cooperation with Trondheim University Hospital, and 30 municipalities in the catchment area of Innlandet Hospital Trust, and Trondheim Municipality. The intervention is developed by an interdisciplinary, experienced research group in close collaboration with user representatives, hospital- and primary health care professionals. It is based on experience, results and preliminary results from foregoing studies by our study group (including NCT03071640 and NCT01742442) and focus group interviews with health professionals.

The design is cluster-randomized, randomizing municipalities and city districts. Patients will be recruited at the radiotherapy units at Innlandet Hospital Trust (primary study center) and Trondheim University Hospital (second study center). Anticipated number of participants from the two hospitals is 102 patients and 60 patients, respectively.

Eligible, consenting patients will be included by the start of radiotherapy (RT), and enter the control or intervention groups in accordance with the assignment of the municipality or city district in which they reside. They will be followed with study specific assessments for one year after end of RT, and for survival for five years.

Assessments:

By the time of inclusion, demographic and medical characteristics (including cancer diagnosis, stage of disease, former and ongoing tumor treatment, ECOG performance status, RT treatment aim (palliative or curative), and comorbidity. Detailed information about the RT schedule will be registered by the end of RT.

Patient reported outcomes (EORTC QLQ-C30 and EQ-5D-5L) will be assessed at baseline, by the end of RT, and thereafter 4, 8, 16, 32 and 52 weeks after RT. Physical performance tests, i.e. Short Physical Performance Battery (SPPB), Timed Up and Go (TUG), grip strength and one-legged balance test, will be applied at baseline and 8 and 16 weeks after the end of RT. Cognitive function will be tested at baseline using the MiniCog.

To evaluate the cost-effectiveness of the intervention in comparison to control (standard care), detailed information on the patients' use of health care services (home based and institutional care) will be registered throughout the intervention period and during follow-up (one year, week 52).

Feasibility will be assessed by a process evaluation, aiming to identify facilitators and barriers for a successful implementation, using mixed methodology. Measures recommended for each patient's intervention plan will be consecutively registered, as will patients' compliance and adherence through weekly contact with the coordinating nurse (log notes). Further data will include interviews with patients and providers. Questionnaires to involved primary health care nurses and other relevant professionals will also be applied.

ELIGIBILITY:
Inclusion Criteria:

* ≥65 years of age
* confirmed cancer diagnosis (histology/cytology)
* living in one of the participating municipalities in the catchment area of Innlandet Hospital Trust or in the municipality of Trondheim
* referred for palliative or curative RT
* fluency in Norwegian, orally and in writing
* ability to fill in self-report questionnaires
* provide written informed consent

Exclusion Criteria:

* severely ill with a life expectancy < 3months
* referred to receive one fraction of RT only (one day treatment)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 178 (Actual)
Dates: Start 2019-05-08 (Actual); Primary Completion 2021-07-25 (Actual); Study Completion 2022-06-10 (Actual)

PRIMARY OUTCOMES:
physical function | 8 weeks following termination of radiotherapy (RT)
  physical function as assessed by patient report using the EORTC QLQ-C30 questionnaire. The analysis will assess the difference between control and intervention groups in physical function measured by the EORTC QLQ-C30 questionnaire at 8 weeks after baseline. Longitudinal analysis of covariance will be performed by estimating a linear mixed model with fixed effects for baseline values, time and interaction between time and group variable. The model will include random effects for patients nested within study cluster.

SECONDARY OUTCOMES:
physical function | trend during follow-up from inclusion to one year after termination of radiotherapy
  physical function as assessed by patient report using the physical function scale from the EORTC QLQ-C30. The scale ranges from 0 (worse) to 100 (best)
global health | 8 weeks after radiotherapy and trend during follow-up from inclusion to one year after radiotherapy
  assessed by the EORTC QLQ-C30 questionnaire's global health/quality of life (QoL) sub-scale (question 29 and 30). The scale ranges from 0 (worse) to 100 (best)
Health related quality of life (HRQoL) | 8 weeks after radiotherapy and trend during follow-up from inclusion to one year after radiotherapy
  assessed by the EQ-5D-5L index values
mobility | 8 weeks after radiotherapy and trend during follow-up from inclusion up to 16 weeks after radiotherapy
  assessed by the short physical performance battery (SPPB)
grip strength | 8 weeks after radiotherapy and trend during follow-up from inclusion up to 16 weeks after radiotherapy
  assessed by dynamometer
the incremental cost-effectiveness ratio (ICER) | 8 weeks after radiotherapy and during follow-up (up to 52 weeks after after radiotherapy)
  We will calculate the intervention cost based on a micro-costing approach. Cost-effectiveness of the intervention will be evaluated by calculating the incremental cost-effectiveness ratio (ICER) that is the difference in mean costs divided by the difference in mean Quality Adjusted Life Years (QALYs). We calculate QALYs by an area under the curve approach under the assumption of piecewise linear change in EQ-5D-5L-index values over time. Missing data will be imputed by multiple imputation and the uncertainty of the ICER will be assessed by performing sensitivity analysis including application of bootstrapping techniques.
Use of health care services | From inclusion through overall follow-up (up to 52 weeks after radiotherapy)
  use of health care services (hospital in- and outpatient services and municipality services in terms of home care, nursing home care and use of other services such as general practitioner, physiotherapist, occupational therapists, and rehabilitation programs)

OTHER OUTCOMES:
mobility | 8 weeks after radiotherapy and trend during follow-up up to 16 weeks after radiotherapy)
  assessed by the Timed Up and Go
balance | 8 weeks after radiotherapy and trend during follow-up up from inclusion to 16 weeks after radiotherapy
  registration of the time the patient is able to maintain balance on one leg
symptom occurence | 8 weeks after radiotherapy and trend during follow-up from inclusion to one year after radiotherapy
  measured by the EORTC QLQ-C30 questionnaire
Body mass index (BMI) | From baseline throughout follow-up up to 52 weeks after RT
  Body mass inndex assessed as weight (kg)/(height m2)
appetite loss (AL) | 8 weeks after radiotherapy and trend during follow-up from inclusion to one year after radiotherapy
  Assessed by the appetite loss subscale on the EORTC QLQ-C30 questionnaire. The scale ranges from 0 (best) to 100 (worse). To be noted is that for all symptom scales of the EORTC QLQ -C30, 0 indicates the best (no symptom), whereas 100 is the worse. This is opposite to the functioning scales such as physical function, global QoL and emotional function
emotional functioning (EF) | 8 weeks after radiotherapy and trend during follow-up from inclusion to one year after radiotherapy
  assessed by the emotional function subscale of theEORTC QLQ-C30 questionnaire. The scale ranges from 0 (worse) to 100 (best)

CONTACTS AND LOCATIONS:
Overall Officials: Marit S Jordhøy, PhD, Principal Investigator — Sykehuset Innlandet HF
Locations (2):
- Norway (2):
  - Innlandet Hospital Trust, Gjøvik
  - St Olav Hospital, Trondheim University Hospital, Trondheim

IPD SHARING:
Plan to Share IPD: No
According to Norwegian Data Protection regulations, sharing of individual participants data is not accepted unless purpose and involved researchers are explicitly stated and approved by the participants (informed consent form) and approved by The Ethical Review Board.

REFERENCES:
- [Background] Royset I, Saltvedt I, Rostoft S, Gronberg BH, Kirkevold O, Oldervoll L, Bye A, Benth JS, Bergh S, Melby L, Halsteinli V, Dohl O, Rostad T, Eriksen GF, Sollid MIV, Rolfson D, Slaaen M. Geriatric assessment with management for older patients with cancer receiving radiotherapy. Protocol of a Norwegian cluster-randomised controlled pilot study. J Geriatr Oncol. 2022 Apr;13(3):363-373. doi: 10.1016/j.jgo.2021.11.001. Epub 2021 Nov 12. PMID 34776384
- [Derived] Sollid MIV, Melby L, Slaaen M, Eilertsen G, Royset IM, Kirkevold O. Experiences With an Intervention Based on Geriatric Assessment With Management: A Qualitative Study. Nurs Open. 2025 Apr;12(4):e70220. doi: 10.1002/nop2.70220. PMID 40223637
- [Derived] Slaaen M, Royset IM, Saltvedt I, Gronberg BH, Halsteinli V, Dohl O, Vossius C, Kirkevold O, Bergh S, Rostoft S, Oldervoll L, Bye A, Melby L, Rosstad T, Eriksen GF, Sollid MIV, Rolfson D, Saltyte Benth J. Geriatric assessment with management for older patients with cancer receiving radiotherapy: a cluster-randomised controlled pilot study. BMC Med. 2024 Jun 10;22(1):232. doi: 10.1186/s12916-024-03446-4. PMID 38853251
- See also: Røyset et al. Protocolpaper, JGO 2022 Apr;13(3):363-373. doi: 10.1016/j.jgo.2021.11.001. — https://pubmed.ncbi.nlm.nih.gov/34776384/

DOCUMENTS (2):
  • Study Protocol (2018-12-09): https://cdn.clinicaltrials.gov/large-docs/37/NCT03881137/Prot_001.pdf
  • Statistical Analysis Plan (2019-03-12): https://cdn.clinicaltrials.gov/large-docs/37/NCT03881137/SAP_000.pdf